CLINICAL TRIAL: NCT06961487
Title: Endovascular Therapy for Large Core Patients With Uncertain Response to Thrombectomy (OUTER LIMITS)
Brief Title: Endovascular Therapy for Large Core Patients With Uncertain Response to Thrombectomy
Acronym: OUTER LIMITS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Gregory W Albers, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 74948
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Acute; Ischemic Stroke, Acute
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Endovascular Thrombectomy (Other): Treatment with one or more thrombectomy devices (only the devices listed in the study protocol are approved for use) plus standard medical therapy for patients with acute ischemic anterior circulation strokes due to large artery occlusion who present with an eligible large ischemic core lesion, and who can be treated within 24 hours of stroke onset.
  Interventions: Procedure: EndovascularThrombectomy; Device: Endovascular thrombectomy with any FDA-approved device
- Medical Management (No Intervention): Standard medical therapy, based on current AHA guidelines

INTERVENTIONS:
Procedure: EndovascularThrombectomy — Endovascular thrombectomy is a minimally invasive procedure that uses catheters and devices to remove blood clots, restoring blood flow to the brain. The procedure involves inserting a catheter (a long, thin tube) into an artery, usually in the groin, and guiding it through the blood vessels to the site of the blocked artery/blood clot in the brain. After the catheter reaches the affected area, a specialized device is guided through the catheter to capture and remove the clot.
  Arms: Endovascular Thrombectomy
Device: Endovascular thrombectomy with any FDA-approved device — The following FDA approved thrombectomy devices will be included:
  Stryker Neurovascular Products:
  * AXS Vecta 74 Aspiration System
  * AXS Vecta Aspiration System (AXS Vecta 71 Aspiration Catheter and AXS Vecta 74 Aspiration Catheter)
  * AXS Vecta Intermediate Catheters (AXS Vecta 71 Intermediate Catheter & AXS Vecta 74 Intermediate Catheter)
  * Trevo XP ProVue Retriever, 3x20 and 4x20
  * Trevo XP ProVue Retriever, 4x30
  * Trevo XP ProVue Retriever, 6x25
  Medtronic Products:
  Solitaire X Revascularization Devices:
  * Solitaire X 4x20, 4x40, 6x40
  * Solitaire X 3x20, 3x40
  Aspiration catheters:
  * React 68
  * React 71
  * REACT-71-115 & REACT-71-125
  MicroVention Inc. Products:
  * SOFIA, Aspiration pump and tubing kit
    * SOFIA Plus Aspiration catheter
  * BOBBY balloon guide catheter
  * ERIC retrieval device
  Other Names: Endovascular Therapy; Endovascular Recanalization Therapy; EVT
  Arms: Endovascular Thrombectomy

SUMMARY:
The purpose of this study is to assess the safety and efficacy of endovascular thrombectomy in both an early and extended time window in patients with large strokes due to large artery occlusion.

DETAILED DESCRIPTION:
This is a pilot prospective randomized trial of patients with acute ischemic anterior circulation strokes due to large artery occlusion who present with an eligible large ischemic core lesion, and who can be treated within 24 hours of stroke onset. The results of this pilot study will be used as preliminary data for a larger NIH-funded multi-center randomized trial to address the knowledge gaps in the management of this patient population.

Eligible patients will be randomized 1:1 to either:

Endovascular therapy plus medical therapy (based on current AHA guidelines)

or

Medical therapy (based on current AHA guidelines)

Endovascular Therapy: Patients randomized to endovascular therapy will be treated with aspiration thrombectomy devices and suction thrombectomy systems approved by the FDA for use in this study. Standard medical therapy, based on current AHA guidelines, will also be provided.

Medical Therapy: Patients randomized to medical therapy will receive standard medical therapy based on current AHA guidelines.

The researchers hope to learn if endovascular therapy plus standard medical therapy in this patient population leads to less disability after stroke than standard medical therapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Signs and symptoms consistent with an acute anterior circulation ischemic stroke and associated brain imaging
2. Baseline NIHSSS is ≥10 and remains ≥10 immediately prior to randomization
3. Treatment can be initiated within 24 hours of stroke onset or time last known well and within 120 minutes of completion of qualifying imaging
4. Functionally independent prior to stroke onset
5. Patient/ Legally Authorized Representative has signed the Informed Consent form.

Exclusion Criteria:

1. Other serious, advanced, or terminal illness (investigator judgment) or life expectancy is less than 6 months.
2. Pre-existing medical, neurological or psychiatric disease that would confound the neurological or functional evaluations
3. Pregnant
4. Unable to undergo a contrast brain perfusion scan with either MRI or CT
5. Known allergy to iodine that precludes an endovascular procedure
6. Treated with tPA or TNK >4.5 hours after time last known well
7. Seizures at stroke onset if it precludes obtaining an accurate baseline NIHSS
8. Baseline blood glucose of <50mg/dL (2.78 mmol) or >400mg/dL (22.20 mmol)
9. Baseline platelet count < 50,000/uL
10. Severe, sustained hypertension (SBP >185 mmHg or DBP >110 mmHg)
11. Current participation in another investigational drug or device study
12. Presumed septic embolus; suspicion of bacterial endocarditis
13. Any other condition that, in the opinion of the investigator, precludes an endovascular procedure or poses a significant hazard to the subject if an endovascular procedure was performed.

NEUROIMAGING Exclusion:

1. Evidence of intracranial tumor (except small meningioma) acute intracranial hemorrhage, neoplasm, or arteriovenous malformation
2. Significant mass effect with midline shift
3. Evidence of internal carotid artery dissection that is flow limiting or aortic dissection
4. Intracranial stent implanted in the same vascular territory that precludes the safe deployment/removal of the neurothrombectomy device
5. Acute symptomatic arterial occlusions in more than one vascular territory confirmed on CTA/MRA (e.g., bilateral MCA occlusions, or an MCA and a basilar artery occlusion).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Disability as measured on the modified Rankin Score | 90 day
  The modified Rankin Scale is a 7 point scale that measures degree of disability after a stroke. The scale range is as follows:
  0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead

SECONDARY OUTCOMES:
Percentage of patients with modified Rankin Scale 0-3 | 90 day
  The modified Rankin Scale is a 7 point scale that measures degree of disability after a stroke. The scale range is as follows:
  0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Percentage of patients requiring hemicraniectomy | from admission to discharge; up to 14 days
  A surgical procedure that involves removing a large bone flap to relieve pressure on the brain due to swelling

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Albers, MD, Principal Investigator — Stanford University; Jeremy Heit, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
we currently do not have a plan to share IPD with other researchers